CLINICAL TRIAL: NCT02001298
Title: The Comparison of the Cardiovascular Effects of Remifentanil and Nitroprusside for Controlled Hypotension
Brief Title: Remifentanil and Nitroprusside for Controlled Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeju National University School of Medicine (Other)
Responsible Party: Principal Investigator, Hyun Jung Kim, Assistant professor, Jeju National University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HJKim3
Record Dates: First submitted 2013-11-24; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Hypotension, Controlled
Keywords: remifentanil; nitroprusside; hypotension
MeSH Terms: conditions — Hypotension | interventions — Remifentanil; Nitroprusside

ARMS (2):
- nitroprusside (Experimental): After induction of anesthesia, controlled hypotension was induced with continuous infusion of nitroprusside. Cardiac index, stroke volume index, and total peripheral resistance index were continuously measured using noninvasive cardiac output monitor (Cheetah NICOM, Cheetah Medical Inc, UK).
  Interventions: Drug: nitroprusside
- remifentanil (Experimental): After induction of anesthesia, controlled hypotension was induced with continuous infusion of remifentanil. Cardiac index, stroke volume index, and total peripheral resistance index were continuously measured using noninvasive cardiac output monitor (Cheetah NICOM, Cheetah Medical Inc, UK).
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil
  Arms: remifentanil
Drug: nitroprusside
  Arms: nitroprusside

SUMMARY:
The purpose of this study is the comparison of the cardiovascular effects of remifentanil and nitroprusside for controlled hypotension

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endoscopic sinus surgery

Exclusion Criteria:

* patient who took any drug to influence this study
* patient with cardiovascular disease, renal disease or liver disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Cardiac index | Cardiac index was continuously measured during controlled hypotension, an average of 90 min
  Cardiac index was continuously measured during controlled hypotension using noninvasive cardiac output monitor. The average of cardiac index during controlled hypotension was compared with baseline value.

SECONDARY OUTCOMES:
Total peripheral resistance index | Total peripheral resistance index was continuously measured during controlled hypotension, an average of 90 min
  Total peripheral resistance index was continuously measured during controlled hypotension using noninvasive cardiac output monitor. The average of total peripheral resistance index during controlled hypotension was compared with baseline value.

OTHER OUTCOMES:
Stroke volume index | Stroke volume index was continuously measured during controlled hypotension, an average of 90 min
  Stroke volume index was continuously measured during controlled hypotension using noninvasive cardiac output monitor. The average of stroke volume index during controlled hypotension was compared with baseline value.

CONTACTS AND LOCATIONS:
Locations (1):
- Jeju National University Hospital, Jeju City, Jeju Special Self-Governing Province, South Korea